CLINICAL TRIAL: NCT04154488
Title: A Phase 1b/2, Open-Label, Multicenter Study of Mavorixafor in Patients With Congenital Neutropenia and Chronic Neutropenia Disorders
Brief Title: A Study of Mavorixafor in Participants With Congenital Neutropenia and Chronic Idiopathic Neutropenia Disorders
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: X4 Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: X4P-001-104
Record Dates: First submitted 2019-11-04; First posted 2019-11-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Neutropenia
Keywords: Chronic congenital neutropenia; Chronic idiopathic neutropenia; SCN; CIN; CXCR4; Mavorixafor; Neutropenia glycogen storage disease type 1b; GSD1b; G6PC3; SLC37A4; GATA2
MeSH Terms: conditions — Neutropenia; Glycogen Storage Disease Id | interventions — mavorixafor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mavorixafor (Experimental): Part 1: Adult participants and adolescent participants who weigh more than 50 kilograms (kg) will receive mavorixafor 400 milligrams (mg) (4 capsules of 100 mg each), orally once on Day 1. Adolescents weighing less than or equal to 50 kg will receive mavorixafor 200 mg (2 capsules of 100 mg each), orally once on Day 1.
  Part 2: Eligible participants from Part 1 will receive once daily dosing of mavorixafor for 6 months.
  Interventions: Drug: Mavorixafor

INTERVENTIONS:
Drug: Mavorixafor — Mavorixafor capsules will be administered per dose and schedule specified in the arm.
  Other Names: X4P-001

SUMMARY:
This is a 2-part study of mavorixafor in participants diagnosed with chronic neutropenia. The main goal of Part 1 (Phase 1b) is to help researchers learn more about how the investigational medicine, mavorixafor, impacts people living with chronic neutropenia (including congenital, idiopathic, and cyclic). In Part 2 (Phase 2), the safety and tolerability of chronic dosing of mavorixafor will be evaluated in a larger participant population and the impact of 6-month chronic dosing of mavorixafor on participant neutropenia.

DETAILED DESCRIPTION:
Part 1: Participants will receive one oral dose of mavorixafor and be monitored for 8 hours to see if neutrophil cell counts increase. Participants screened after implementation of Protocol Version 8.0, do not need to enter Part 1 and can start with the Part 2 Screening visit (Day -28 to Day -1).

Part 2: For participants enrolled in the study before implementation of Protocol Version 8.0, Part 2 will include those who completed Part 1 and exhibited a response to treatment. Eligible participants from Part 1 enrolled in the study before implementation of Protocol Version 8.0, can directly roll-over to the Baseline (Day -3 to Day -1) visit in Part 2. Participants will receive once daily oral dosing of mavorixafor for 6 months and be monitored throughout to see if neutrophil cell counts increase.

Study visits can be conducted at-home or at one of many study clinic locations, depending on the participant's preference.

ELIGIBILITY:
Key Inclusion Criteria:

For all participants (Parts 1 and 2):

* Sign the informed consent form (ICF) and be willing and able to comply with the protocol.
* Weigh ≥15 kg
* Agree to use a highly effective form of contraception if sexually active.
* Participants may be eligible for the study whether they are on or off granulocyte-colony stimulating factor (G-CSF) treatment.

  * Note: Participants who are on G-CSF must be on a stable dose for ≥14 days prior to the Baseline visit and should not have an ANC ≥10,000 cells/μL.
  * Note: Participants who are not on G-CSF must be off for ≥14 days prior to the Baseline visit and have an ANC ≤1000 cells/µL at the Screening visit.
  * Note: Participants with Shwachman-Diamond syndrome, Cohensyndrome, and warts, hypogammaglobulinemia, infections and myelokathexis syndrome are eligible. Other types of chronic neutropenic disorders may also be eligible for enrollment upon discussion and approval with Sponsor and Study Medical Monitor.
* Have been diagnosed with chronic neutropenia for ≥6 months prior to the Screening visit that is not attributable to medications, active or recent (≤3 months) infections, or malignant cause.

Part 2 only:

* Participants enrolled in the study before implementation of Protocol Version 8.0 must have completed Part 1 and exhibited a positive response to treatment.
* Participant has a history of symptomatic chronic neutropenia confirmed by the Investigator.

Key Exclusion Criteria (Parts 1 and 2):

* Known systemic hypersensitivity to the mavorixafor drug substance or its inactive ingredients.
* Is pregnant, breastfeeding, or plans to become pregnant over the next 8 months.
* Known history of a positive serology or viral load for human immunodeficiency virus (HIV) or a known history of acquired immune deficiency syndrome.
* Known active SARS-CoV-2 virus (COVID-19) infection or a positive test within the local accepted clinical and governmental guidelines for a communicable window.
* At the Screening Visit, has laboratory test results meeting one or more of the following criteria:

  * Positive hepatitis C virus (HCV) antibodies with confirmation by HCV-ribonucleic acid polymerase chain reaction reflex testing.
  * Positive hepatitis B surface antigen (hBsAg) or hepatitis B core antibody (hBcAb).
  * Note: If a participant tests negative for hBsAg but positive for hBcAb, the participant would be considered eligible if the participant tests positive for antibody to hBsAg reflex testing.
* At the Screening visit, has laboratory test results meeting one or more of the following criteria:

  * Hemoglobin <9.0 grams/deciliter (g/dL)
  * Platelets <30,000/μL
  * Estimated glomerular filtration rate (eGFR) ≤60 mL/minute/1.73 meter (m)^2, as estimated by the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation
  * Serum aspartate transaminase >2.5 x upper limit of normal (ULN)
  * Serum alanine transaminase >2.5 x ULN
  * Total bilirubin >1.5 x ULN (unless due to Gilbert's syndrome, in which case total bilirubin greater than or equal to (≥) 3.0 x ULN and direct bilirubin >1.5 x ULN)
* ≤14 days before Day 1, received any of the following treatments:

  * Systemic glucocorticoids (>5 mg prednisone equivalent per day).
  * Medication prohibited based on cytochrome P450 (CYP)2D6 potential for interaction.
* Is taking a medication which is a strong inhibitor of CYP3A4, unless the Investigator and Medical Monitor conclude that the medication must be used during the study and is permissible with modification of mavorixafor dose.
* Has an infection requiring use of systemic antibiotics ≤4 weeks before the Baseline visit.
* Has a medical or personal condition that may potentially compromise the safety or compliance of the participant, or may preclude the participant's successful completion of the clinical study or that in the opinion of the Investigator or the Sponsor could interfere with the objectives of the study.
* Has had major surgery ≤4 weeks before the Baseline visit.
* Inability to ingest mavorixafor capsules.
* Has an active malignancy or history of (≤5 years prior to enrollment) in the study of solid, metastatic, or hematologic malignancy. Exception: basal cell carcinoma in situ of the skin that has been adequately treated.
* Diagnosed or has suspected congenital long QT syndrome. Any history of clinically significant ventricular arrhythmias (such as ventricular tachycardia, ventricular fibrillation, or torsades de pointes); any history of arrhythmia will be discussed with the sponsor's medical monitor before participant's entry into the study.
* Prolonged corrected QT interval using Fridericia's formula at the Screening visit electrocardiogram (ECG) (>450 milliseconds [ms])

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-10-16 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) After a Single Dose of Mavorixafor | Baseline through Day 1 and 7 days follow-up
Number of Participants With Treatment-Emergent Adverse Events (TEAEs) After Multiple Doses of Mavorixafor | Baseline through Month 6 and 30 days follow-up
Change From Baseline in Absolute Neutrophil Count (ANC) to 8 hours Post-dose On Day 1 | Baseline, 8 hours Post-dose On Day 1
Change From Baseline in ANC to Month 6 | Baseline, Month 6

SECONDARY OUTCOMES:
Serum Concentration of Mavorixafor in Relation to ANC and Area Under the Curve (AUC) for ANC (AUCANC) | 0 (pre-dose), 60 minutes and 2, 3, 4, 6, and 8 hours post-dose on Day 1
Serum Concentrations of Mavorixafor | 0 (pre-dose) up to Month 6
Change from Baseline in Absolute Lymphocyte Count (ALC) | Baseline, Month 6
Change from Baseline in Total White Blood Cells (WBC) | Baseline, Month 6
Change from Baseline in Absolute Monocyte (AMC) | Baseline, Month 6
AUC of ANC (AUCANC) | Baseline up to Month 6
AUC of ALC (AUCALC) | Baseline up to Month 6
AUC of AMC (AUCAMC) | Baseline up to Month 6
AUC of WBC (AUCWBC) | Baseline up to Month 6

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - USF Health Department of Pediatrics, St. Petersburg, Florida
  - University of Iowa Hospital and Clinics, Iowa City, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Texas, Southwestern, Dallas, Texas
  - University of Washington, Seattle, Washington